CLINICAL TRIAL: NCT00754871
Title: A Double-blind, Randomized, Dose-controlled Study to Evaluate Pharmacodynamic Properties of Four Oral Doses of Dienogest (DNG) in 100 Healthy Young Female Volunteers Over a Period of Two Cycles up to a Maximum of 72 Days
Brief Title: Pharmacodynamic Characterization of Dienogest
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 13180; 2008-003611-13 (EudraCT Number)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Pharmacodynamics
MeSH Terms: interventions — dienogest

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Dienogest (81150037)
- Arm 2 (Experimental)
  Interventions: Drug: Dienogest (81150231)
- Arm 3 (Experimental)
  Interventions: Drug: Dienogest (SH T00660A)
- Arm 4 (Experimental)
  Interventions: Drug: Dienogest (81150746)

INTERVENTIONS:
Drug: Dienogest (81150037) — daily oral intake of 0.5 mg dienogest over two cycles or a max. of 72 days
  Arms: Arm 1
Drug: Dienogest (81150231) — daily oral intake of 1.0 mg dienogest over two cycles or a max. of 72 days
  Arms: Arm 2
Drug: Dienogest (SH T00660A) — daily oral intake of 2.0 mg dienogest over two cycles or a max. of 72 days
  Arms: Arm 3
Drug: Dienogest (81150746) — daily oral intake of 3.0 mg dienogest over two cycles or a max. of 72 days
  Arms: Arm 4

SUMMARY:
This study will be investigated what mechanism of action Dienogest has. The growth of the follicles, the endometrium, the hormones in the blood and the mucus that is produced by the cervix that will be looked upon. Four different dosages of Dienogest (0.5 mg, 1 mg, 2 mg and 3 mg) will be investigated in healthy young women over two cycles, or up to a maximum of 72 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body-Mass-Index (BMI): 18 - 30 kg/m²
* Healthy female volunteers
* Age 18-35 years (smoker not older than 30 years, inclusive)
* At least 3 months since delivery, abortion or lactation
* Willingness to use non-hormonal methods of contraception during entire study

Exclusion Criteria:

* Contraindications for use of progesterone-only pills or combined oral contraceptives (e.g. history of venous/arterial thromboembolic disease)
* Use of systemic or topical medications or substances which oppose the study objectives or which might influence them within 4 weeks prior to start of the pre-treatment cycle
* Clinically relevant findings (blood pressure, physical and gynecological examination, laboratory examination)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
No primary variables defined, all variables are considered exploratory since no confirmatory statistical analysis planned | No primary variables defined, all variables are considered exploratory since no confirmatory statistical analysis planned

SECONDARY OUTCOMES:
Course of gonadotropins (FSH, LH, P, E2) | During pre-treatment and treatment cycles (3 months)
Endometrial thickness | During pre-treatment and treatment cycles (3 months)
Grading of ovarian activity | During pre-treatment and treatment cycles (3 months)
Effects on the cervix and the cervical mucus | During pre-treatment and treatment cycles (3 months)
mRNA expression profile of endometrial biopsies and in blood | once in pre-treatment and during treatment
Concentrations of DNG in serum | During pre-treatment and treatment cycles (3 months)
Safety and tolerability | During pre-treatment and treatment cycles (3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Groningen, Netherlands

REFERENCES:
- [Result] Klipping C, Duijkers I, Remmers A, Faustmann T, Zurth C, Klein S, Schuett B. Ovulation-inhibiting effects of dienogest in a randomized, dose-controlled pharmacodynamic trial of healthy women. J Clin Pharmacol. 2012 Nov;52(11):1704-13. doi: 10.1177/0091270011423664. Epub 2011 Nov 29. PMID 22128200
- See also: Click here and search for product information by EMA — http://www.clinicaltrialsregister.eu